CLINICAL TRIAL: NCT01410656
Title: Prostate Cancer Survivors MOving Toward Exercise (PROMOTE) Trial
Acronym: PROMOTE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Principal Investigator, Kerry Courneya, Professor, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RES-0006611
Record Dates: First submitted 2011-07-19; First posted 2011-08-05 (Estimated); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Prostate Cancer
Keywords: Survivors
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard PA Recommendation (No Intervention): Received the standard physical activity recommendation.
- Telephone Implementation Intention (Experimental): Behavioural Telephone Assisted Implementation Intention Intervention
  Interventions: Behavioral: Telephone Implementation Intention
- Self-completed implementation intention (Experimental): Self-administered implementation intention intervention.
  Interventions: Behavioral: Self-completed implementation intention

INTERVENTIONS:
Behavioral: Telephone Implementation Intention — Telephone implementation intention counseling
  Arms: Telephone Implementation Intention
Behavioral: Self-completed implementation intention — Self-administered implementation intention intervention
  Arms: Self-completed implementation intention

SUMMARY:
The primary purpose of the study is to determine the effects of an implementation intention intervention on physical activity (PA) behaviour in prostate cancer survivors. Secondary aims are to (a) compare the effects of a telephone-assisted implementation intention intervention against a self-administered implementation intention intervention and a standard recommendation group on physical activity behaviour and (b) document the effects of these interventions on quality of life (QoL), fatigue, symptom management, and physical functioning.

Hypotheses: Evidence exists that an implementation intention intervention can lead to significant improvements in PA levels and that regular PA has been shown to improve QoL, fatigue levels, manage symptoms and improve physical functioning in cancer survivors'. As such, the following hypotheses were generated: (1) prostate cancer survivors exposed to the researcher-assisted implementation intention intervention will have higher PA levels at the 1- and 3-month follow-ups compared to the self-completed implementation intention intervention and the standard recommendation group; (2) prostate cancer survivors in the researcher-assisted implementation intention intervention will show significant improvements in QoL, fatigue levels, symptom management, and physical functioning compared to the self-completed implementation intention intervention and the standard recommendation group at the 1- and 3-month follow-up; and (3) prostate cancer survivors in the self-completed implementation intention intervention will have higher PA levels, and better improvements in QoL, fatigue levels, symptom management, and physical functioning compared to the standard recommendation group at the 1- and 3-month follow-ups.

DETAILED DESCRIPTION:
BACKGROUND:

Prostate cancer remains the most frequently diagnosed cancer among Canadian men, with an estimated 24,600 men being diagnosed in 2010. In Alberta specifically, roughly 2,500 men will be diagnosed with prostate cancer, and 440 men will die of the disease in 2010 (Canadian Cancer Society, 2011). Improvements in the treatment of prostate cancer has reduced tumour growth and improved survival rates, however, it has also been associated with significant negative changes in cancer survivors' quality of life, physical functioning, body fat percentage and fatigue levels that may persist for years following treatment. One behavioural strategy that has been consistently shown to combat these negative side effects and enhance psychosocial and physical well-being in prostate cancer survivors is physical activity. Unfortunately it has been established that physical activity levels decline significantly from pre-diagnosis to during treatment and may never regain pre-diagnosis levels; thus it is important to test novel, innovative and inexpensive ways to increase physical activity patterns in prostate cancer survivors.

PURPOSE:

The primary purpose of the study is to determine the effects of an implementation intention intervention on physical activity behaviour in prostate cancer survivors. Secondary aims are to (a) compare the effects of a telephone-assisted implementation intention intervention against a self-administered implementation intention intervention and a standard recommendation group on physical activity behaviour and (b) document the effects of these interventions on quality of life, fatigue, symptom management, and physical functioning.

METHODS:

A three-arm randomized controlled trial for prostate cancer survivors will be performed through the Alberta Cancer Registry. To obtain a sample of at least 300 participants, 1500 prostate cancer survivors will be contacted in the initial mail-out. Following the initial mail-out prostate cancer survivors agreeing to participate in the study will be randomized to one of the three conditions. All groups will receive a written physical activity recommendation, as well as the 2008 Physical Activity Guidelines. In addition to the physical activity materials, participants in the telephone-assisted and self-administered groups will be asked to complete an implementation intention intervention. Finally, the telephone-assisted group will receive a 10-20 minute telephone call to assist them with the completion of implementation intention intervention. Measures at baseline (i.e., initial mail-out) will include self-reported physical activity, demographic, health and medical factors, quality of life, fatigue, physical functioning. Follow-up at month 1 and 3 following the intervention will include self-reported physical activity, quality of life, fatigue and physical function measures.

SUMMARY:

This mail-out study will offer insight into the effects of an implementation intention intervention on physical activity levels in an understudied cancer population, and further explore the effect of physical activity as part of the usual care recommended for the treatment of prostate cancer on quality of life, fatigue and symptom management.

ELIGIBILITY:
Inclusion Criteria:

* Prostate cancer survivors
* at least 18 years old
* proficient in English

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 423 (Actual)
Dates: Start 2011-05; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Change in Physical activity Levels From Baseline to Month 1 and Month 3 | baseline, 1 month, 3 months
  Measured by the Leisure score index. Looking for change in Physical Activity levels from baseline to month 1 and month 3 follow-ups.

SECONDARY OUTCOMES:
Quality of life/ physical functioning | baseline, 3 months
  Looking for change in the FACT-P and SF-36.
fatigue | baseline, 3 months
  Looking for change in the FACIT-F

CONTACTS AND LOCATIONS:
Overall Officials: Kerry S Courneya, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

REFERENCES:
- [Derived] McGowan EL, Fuller D, Cutumisu N, North S, Courneya KS. The role of the built environment in a randomized controlled trial to increase physical activity among men with prostate cancer: the PROMOTE trial. Support Care Cancer. 2017 Oct;25(10):2993-2996. doi: 10.1007/s00520-017-3798-1. Epub 2017 Jun 27. PMID 28656468
- [Derived] McGowan EL, North S, Courneya KS. Randomized controlled trial of a behavior change intervention to increase physical activity and quality of life in prostate cancer survivors. Ann Behav Med. 2013 Dec;46(3):382-93. doi: 10.1007/s12160-013-9519-1. PMID 23783829